CLINICAL TRIAL: NCT03938181
Title: Influence of Preoperative Fluid Intake on the Onset of Postoperative Acute Kidney Injury in Cardiac Surgery Patients: the HYDRATE-CSX Trial
Brief Title: Influence of Preoperative Fluid Intake on the Onset of Postoperative Acute Kidney Injury
Acronym: HYDRATE-CSX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 3CARE_BOÄ_18-004_Hydrate-CSX
Record Dates: First submitted 2019-05-02; First posted 2019-05-06 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Thoracic Surgery; Acute Kidney Injury; Critical Care
Keywords: cardiac surgery patients; acute renal failure; intensive care
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the influence of preoperative fluid and food intake in cardiac surgery patients on the development of postoperative AKI.

DETAILED DESCRIPTION:
Acute renal failure (ARF) and the need for renal replacement therapy (RRT) is a major complication after cardiac surgery, associated with mortality and an increased risk to develop end-stage renal disease. Cardiac surgery patients are at increased risk to develop acute kidney failure due to ischaemia-reperfusion injury, cardiopulmonary bypass (CPB) induced inflammation and haemolysis, hemodynamic alterations, vasoconstriction and resulting reduced renal perfusion. According to the current literature, AKI occurs in average in 20-30% after cardiac surgery with an incidence of RRT in 1-5%. Several reviews revealed the literature and concluded that , inter alia, euvolemia, adequate nutrition, the avoidance of nephrotoxic drugs and anemia optimization belong to the most effective prevention strategies.

Patients are instructed to follow the nil per os (NPO) guidelines, including abstinence of clear liquids for >2 hours preoperative as well as fasting time of light foods for > 6 hours and fatty foods for >8 hours prior to surgery. However, these guidelines encourage patients to continue PO hydration until 2 h before surgery in order to optimize the volume status. Besides the fact that NPO lasts in average critically longer than required, surgery delay is a common issue and may lead to an exceedance of NPO up to twice as long as required.

Data about the exact mechanism is still sparse, but preoperative iv hydration may correct or even expand intravascular volume, improve renal perfusion and induce diuresis, stimulate endogenous natriuretic peptides release and inactivate the renin-angiotensin-aldosterone system (RAAS).

Large trials on this very relevant topic in these high risk cardiac surgery patients are absolutely missing. Therefore, this prospective observational study aims to investigate the influence of varied preoperative fluid and food intake in cardiac surgery patients on the development of postoperative AKI.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age) scheduled to undergo elective cardiac surgery with the use of cardiopulmonary bypass (CPB) and cardioplegic arrest

Exclusion Criteria:

* Patients not willing to participate or not able to give informed consent
* Patients receiving contrast agents within 72 hours before surgery
* Patients with preoperative need for renal replacement therapy
* Patients receiving an extracorporeal mechanical assist device (e.g. ECLS) or for advanced heart failure therapies (e.g. TAH, VAD) will be excluded.
* Patients participating in another interventional trial
* Pregnant or lactating patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective cardiac surgery at the University Hospital RWTH Aachen
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2020-01-15 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Acute kidney injury | 30 days
  Acute kidney injury
Renal replacement therapy | 7 days postoperative
  Renal replacement therapy
Kidney-failure-free days | 7 days postoperative
  defined as the number of days in which a patient had no acute kidney injury and no need for RRT

SECONDARY OUTCOMES:
Major Adverse Kidney Events | 30 days
  death, dialysis or persistent renal dysfunction
Fluid intake since hospital admission until surgery (ml/h) | 30 days
  Fluid intake since hospital admission until surgery (ml/h)
Calorie intake since hospital admission (kcal/d) | 30 days
  Calorie intake since hospital admission (kcal/d)
Preoperative abstinence of fluids (minutes) | 30 days
  Preoperative abstinence of fluids (minutes)
Preoperative abstinence of food (minutes) | 30 days
  Preoperative abstinence of food (minutes)
ICU length of stay (hours) | 30 days
  ICU length of stay (hours)
Hospital length of stay since surgery (days) | 30 days
  Hospital length of stay since surgery (days)
Mortality until hospital discharge/ 30 days | up to 30 days
  Mortality until hospital discharge/ 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Julia Ney, Dr. med., Principal Investigator — RWTH Aachen University
Locations (1):
- University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No